CLINICAL TRIAL: NCT04086108
Title: Plasmakinetics of GABA From Tomatoes as Compared to GABA From a Supplement, After a Single Oral Administration in Healthy Young Men
Brief Title: Relative Oral Bioavailability of GABA From Tomatoes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Nunhems (Unknown); Agrico Research (Unknown); Avebe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19/13
Record Dates: First submitted 2019-06-18; First posted 2019-09-11 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: GABA Plasmakinetics
Keywords: GABA; Glutamate; Tomato; Plasmakinetics; Bioavailability
MeSH Terms: interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Intervention Model Description: For the study, research subjects will visit the university on four test days separated by a wash out period of one week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tomato (Experimental): Single oral administration
  Interventions: Dietary Supplement: Tomato
- GABA supplement (Experimental): Single oral administration
  Interventions: Dietary Supplement: GABA supplement
- Glutamate supplement (Experimental): Single oral administration
  Interventions: Dietary Supplement: Glutamate supplement
- Placebo (No Intervention): Single oral administration, same volume of water that is distributed in the other arms

INTERVENTIONS:
Dietary Supplement: Tomato — A maximum of 1 kilo pureed tomatoes, containing 1 gram of GABA.
  Arms: Tomato
Dietary Supplement: GABA supplement — 1 gram of GABA dissolved in water.
  Other Names: Gamma-aminobutyric acid
  Arms: GABA supplement
Dietary Supplement: Glutamate supplement — A maximum of 8 grams glutamate, adjusted to amount of glutamate given in the tomato arm. Dissolved in water.
  Arms: Glutamate supplement

SUMMARY:
In this four-way crossover study, a plasmakinetic profile of GABA from tomatoes as compared to a gamma-aminobutyric acid (GABA) supplement in healthy young men will be established. In addition, a plasmakinetic profiles of glutamate from a supplement and from tomatoes as well as the effects of glutamate from tomatoes and a supplement on the GABA plasma levels will be determined. This study will therefore provide information about the effect of a food matrix on GABA plasmakinetics.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 25 kg/m2
* Age is between 18 and 28 years
* Good general health
* Male
* Veins suitable for blood sampling
* Able to speak Dutch

Exclusion Criteria:

* Is currently suffering from a disease including mental disorders
* Has had any gastrointestinal condition/disease within the 3 months prior to the intervention
* Haemoglobin (Hb) level < 8.5 mmol/L
* Has used medication in the two months before and/or during the intervention. Occasional use of NSAIDs or paracetamol (<once a week on average) are is allowed.
* Reported weight loss or weight gain of > 2 kg in the month prior to the intervention
* Use of dietary supplements, 3 weeks before-, or during the intervention.
* Allergic to products that are provided as part of the standardised diet
* Unwilling to consume the products that are part of the standardised diet
* Allergic to tomatoes
* (History of) drug abuse, in this case meaning >1 x per month use of recreational drugs
* Smoking
* Alcohol consumption of >10 standardised glasses per week.
* Not able to refrain from alcohol consumption 2 days before each test day
* Recent or planned blood donation (<3 month prior to first study day or during intervention)
* Personnel of Wageningen University, department of Human Nutrition and Health,
* Currently participating in other research or was participating in another study within 1 month of the intervention or within 3 months if invasive procedures were used.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC ) of plasma-time curves of GABA | 6 months
  After intake of a GABA supplement and tomatoes.
Peak Plasma Concentration (Cmax) of plasma-time curves of GABA | 6 months
  After intake of a GABA supplement and tomatoes.
Time to Peak Plasma Concentration (Tmax) of plasma-time curves of GABA | 6 months
  After intake of a GABA supplement and tomatoes.
Half-life (T1/2) of plasma-time curves of GABA | 6 months
  After intake of a GABA supplement and tomatoes.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of plasma-time curves of glutamate | 6 months
  After intake of a glutamate supplement and tomatoes
Peak Plasma Concentration (Cmax) of plasma-time curves of glutamate | 6 months
  After intake of a glutamate supplement and tomatoes
Time to Peak Plasma Concentration (Tmax) of plasma-time curves of glutamate | 6 months
  After intake of a glutamate supplement and tomatoes
Half-life (T1/2) of plasma-time curves of glutamate | 6 months
  After intake of a glutamate supplement and tomatoes
Area under the plasma concentration versus time curve (AUC) AUC of plasma-time curves of GABA in response to a glutamate supplement. | 6 months
  This will be compared to the plasma time-curves of GABA after tomato intake.
Peak Plasma Concentration (Cmax) of plasma-time curves of GABA in response to a glutamate supplement. | 6 months
  This will be compared to the plasma time-curves of GABA after tomato intake.
Time to Peak Plasma Concentration (Tmax) of plasma-time curves of GABA in response to a glutamate supplement. | 6 months
  This will be compared to the plasma time-curves of GABA after tomato intake.
Half-life (T1/2) of plasma-time curves of GABA in response to a glutamate supplement. | 6 months
  This will be compared to the plasma time-curves of GABA after tomato intake.

CONTACTS AND LOCATIONS:
Overall Officials: Renger Witkamp, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Bie TH, Balvers MGJ, de Vos RCH, Witkamp RF, Jongsma MA. The influence of a tomato food matrix on the bioavailability and plasma kinetics of oral gamma-aminobutyric acid (GABA) and its precursor glutamate in healthy men. Food Funct. 2022 Aug 15;13(16):8399-8410. doi: 10.1039/d2fo01358d. PMID 35852458